CLINICAL TRIAL: NCT01546207
Title: Stepwise Approach To sUbstrate Modification for Ventricular Tachycardia
Acronym: STRATUM VT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment
Sponsor: Vivek Reddy (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Director Cardiac Arrhythmia Service, Professor of Medicine, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 12-0045
Record Dates: First submitted 2012-02-13; First posted 2012-03-07 (Estimated); Results first posted 2014-04-24 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Ventricular Tachycardia; Catheter Ablation; Tachycardia, Ventricular
Keywords: ventricular tachycardia; catheter ablation; VT
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- catheter-based ablation (Other): catheter ablation - a medical procedure used to treat some types of arrhythmia
  Interventions: Procedure: catheter-based ablation

INTERVENTIONS:
Procedure: catheter-based ablation — specific electrophysiological and mapping techniques of activation and entrainment mapping during ongoing VT. Substrate mapping and ablation (substrate modification.) catheter ablation - a medical procedure used to treat some types of arrhythmia

SUMMARY:
The goal of this trial is to test the impact of a step-wise approach for catheter ablation of recurrent ventricular tachycardia, (irregular heart rhythms that originate in the bottom chambers of the heart), in patients with a previous heart attack for whom catheter ablation is clinically indicated.

DETAILED DESCRIPTION:
Sudden cardiac death due to VT (ventricular tachycardia) or VF (ventricular fibrillation) occurs at an estimated rate of 300,000 events per year in United States, accounting for 5.6% of annual mortality22. A significant proportion of patients treated with ICDs (implantable defibrillators) will receive shocks due to recurrent VT, resulting in increased mortality8. As a result, catheter-based ablation has emerged as an effective treatment for recurrent VT. However, no study has assessed the impact of a step-wise approach on the outcome of catheter ablation of VT. The investigators propose a prospective, multicenter, non-randomized, single-arm trial to evaluate the impact of a step-wise approach to catheter ablation on ventricular tachycardia recurrence. Given the increasing use of catheter ablation in patients with recurrent ventricular tachycardia, this study will answer a critical question regarding the impact of a step-wise approach on the inducibility of VT at the end of the procedure and clinical recurrences of ventricular arrhythmias at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 90 years.
* History of coronary artery disease.
* Presence of, or planned for, an ICD prior to discharge.
* Presentation for management of ICD shock/ATP therapy or monomorphic ventricular tachycardia.

Exclusion Criteria:

* Ventricular arrhythmia not thought to be due to CAD.
* Unstable angina
* CVA within 30 days.
* Protruding left ventricular thrombus or critical aortic stenosis on pre-ablation echocardiography
* Pregnancy
* Any condition resulting in an absolute contraindication to anticoagulation
* Inability to follow-up at ICD clinic.
* Inability to give informed consent.
* Non-inducible for sustained monomorphic ventricular tachycardia.
* Prior substrate guided ablation.
* Definite need for epicardial ablation, as determined by the primary operator.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (10):
- United States (6):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Loyola University, Maywood, Illinois
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel-Deaconess Medical Center, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Hospital Regional Sao Jose, Santa Catarina, Brazil
- Southlake Regional Health Center, Newmarket, Ontario, Canada
- Homolka Hospital, Prague, Czechia
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 12/2011 to 7/2013, at a medical clinic at MSSM.
Period: Overall Study
Arm/Group | Catheter-based Ablation
Started | 4
Completed | 3
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Catheter-based Ablation
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.75 (7.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Catheter Ablation
Description: The procedural efficacy as defined as acute success of a standardized step-wise approach for substrate-based catheter ablation of recurrent ventricular tachycardia in patients with coronary artery disease and prior ventricular tachycardia or appropriate therapy. Acute success will be defined as the ability to render VT non-inducible with a standardized complete stimulation protocol. catheter ablation - a medical procedure used to treat some types of arrhythmia
Time Frame: at time of catheter ablation procedure (intraoperative)
Population: Given the small sample size, we did not analyze the data as there would be no statistical significance.
Arm/Group | Catheter-based Ablation
Number analyzed (Participants) | 0

2. Secondary Outcome: ICD Interrogation
Description: Chronic success will be defined as no recurrence of sustained VT or VT resulting in ICD therapies (ATP and/or ICD shocks) at 6 months follow-up as compared to baseline.
Time Frame: baseline and 6 months follow-up
Reporting Status: Not Posted

3. Secondary Outcome: Procedural Safety
Description: 2) Procedural safety as defined by the number of complication within 1week associated with the procedure.
Time Frame: 1 week post-op
Reporting Status: Not Posted

4. Secondary Outcome: Signal-Average ECG
Description: Relationship between change in pre/post saECG and success of the step-wise ablation strategy
Time Frame: baseline and post-op day one after procedure
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Catheter-based Ablation
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheter-based Ablation (N=4)
Ventricular Tachycardia (Cardiac disorders) | 1 (4)
pseudoaneurysm with hematoma (Blood and lymphatic system disorders) | 1 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheter-based Ablation (N=4)
hematuria (Renal and urinary disorders) | 1 (1)
pericardial effusion (Cardiac disorders) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (1)
sustained Ventricular Tachycardia (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to poor enrollment. Data analysis not done - there is not enough data for meaningful analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes